CLINICAL TRIAL: NCT02964273
Title: A Phase 3b, Two-part, Multicenter, One Year Randomized, Double-blind, Placebo-controlled Trial of the Safety, Pharmacokinetics, Tolerability, and Efficacy of Tolvaptan Followed by a Two Year Open-label Extension in Children and Adolescent Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: Safety, Pharmacokinetics, Tolerability and Efficacy of Tolvaptan in Children and Adolescents With ADPKD (Autosomal Dominant Polycystic Kidney Disease)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 156-12-298; 2016-000187-42 (EudraCT Number)
Record Dates: First submitted 2016-09-15; First posted 2016-11-16 (Estimated); Results first posted 2023-01-03 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: Autosomal Dominant Polycystic Kidney Disease; ADPKD; Tolvaptan; Renal cysts; Chronic Kidney Disease; Genetic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Renal Insufficiency, Chronic | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase A: Tolvaptan (Experimental): Participants received tolvaptan tablets, orally as a split dose (with the first dose taken upon awakening and the second dose taken approximately 8 hours later), and starting doses based on their weight as per the following specifications: ≥20 to 45 kg: 15/7.5 mg; ≥45 to ≤75 kg: 30/15 mg; >75 kg: 45/15 mg, for 1 week. The starting dose was up-titrated (≥20 to <45 kg: 30/15 mg; ≥45 to ≤75 kg: 45/15 mg; >75 kg: 60/30 mg) after 1 week based upon tolerability and thereafter participants continued the same dose for 12 months. Doses may be titrated down dependent upon participant tolerability.
  Interventions: Drug: Tolvaptan
- Phase A: Placebo (Placebo Comparator): Participants received matching-placebo tablets, orally as a split-dose (with the first dose taken upon awakening and second dose taken approximately 8 hours later), and starting dose based on their weight as per the following specifications: ≥20 to <45 kg: 15/7.5 mg; ≥45 to ≤75 kg: 30/15 mg; >75 kg: 45/15 mg, for 1 week. The starting dose was up-titrated (≥20 to <45 kg: 30/15 mg; ≥45 to ≤75 kg: 45/15 mg; >75 kg: 60/30 mg) after 1 week based upon tolerability and thereafter participants continued the same dose for 12 months. Doses may be titrated down dependent upon participant tolerability.
  Interventions: Drug: Tolvaptan Matching-placebo
- Phase B: Prior Tolvaptan (Experimental): Qualified participants (defined as those who were willing to continue in the trial and who did not have any adverse events [AEs] that would require investigational medicinal product [IMP] discontinuation) who received tolvaptan and completed Phase A were enrolled in Phase B and received tolvaptan tablets, orally as a split dose (with the first dose taken upon awakening and the second dose taken approximately 8 hours later), and starting dose based on their body weight as per following specifications: ≥20 to <45 kg: 15/7.5 mg; ≥45 to ≤75 kg: 30/15 mg; >75 kg: 45/15 mg, for 1 week. The starting dose was up-titrated (≥20 to <45 kg: 30/15 mg; ≥45 to ≤75 kg: 45/15 mg; >75 kg: 60/30 mg) after 1 week based upon tolerability and thereafter participants continued the same dose for 24 months. Doses may be titrated down dependent upon participant tolerability.
  Interventions: Drug: Tolvaptan
- Phase B: Prior Placebo (Experimental): Qualified participants (defined as those who were willing to continue in the trial and who did not have any AEs that would require IMP discontinuation) who received matching-placebo and completed Phase A, were enrolled in Phase B and received tolvaptan tablets, orally as a split dose (with the first dose taken upon awakening and the second dose taken approximately 8 hours later), based on their current body weight as per following specifications: ≥20 to <45 kg: 15/7.5 mg; ≥45 to ≤75 kg: 30/15 mg; >75 kg: 45/15 mg, for 1 week. The starting dose was up-titrated (≥20 to <45 kg: 30/15 mg; ≥45 to ≤75 kg: 45/15 mg; >75 kg: 60/30 mg) after 1 week based upon tolerability and thereafter participants continued the same dose for 24 months. Doses may be titrated down dependent upon participant tolerability.
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan spray-dried, immediate release tablets
  Other Names: OPC-41061
  Arms: Phase A: Tolvaptan; Phase B: Prior Placebo; Phase B: Prior Tolvaptan
Drug: Tolvaptan Matching-placebo — Tolvaptan matching-placebo tablets
  Arms: Phase A: Placebo

SUMMARY:
The primary objective of the study is to assess the long term safety of treatment with tolvaptan in children and adolescents with autosomal dominant polycystic kidney disease (ADPKD). The secondary objective is to assess the pharmacodynamics, pharmacokinetics, and efficacy of tolvaptan in the same participant population.

DETAILED DESCRIPTION:
Tolvaptan has been demonstrated to delay the decline of kidney function in adults with rapidly progressing ADPKD (chronic kidney disease [CKD] stages 1 to 3) as measured by estimated glomerular filtration rate (eGFR) and Total Kidney Volume (TKV).

This trial will be the first trial of tolvaptan in children and adolescents with ADPKD.

Participants in this study will be randomly assigned to one of two groups in Phase A; tolvaptan or placebo. Participants will have an equal chance of being assigned to either treatment group and will be stratified by age and gender into the following cohorts:

* Female participant ages 12 to 14 years, inclusive
* Female participant ages 15 to 17 years, inclusive
* Male participant ages 12 to 14 years, inclusive
* Male participant ages 15 to 17 years, inclusive

Phase (A) of this study will last 12 months. After that time, all participants who qualify will be assigned tolvaptan and will be treated with tolvaptan for 24 months (Phase B).

A qualified participant is defined as one who has completed Phase A on investigational medicinal product (IMP), is willing to continue in the trial, and who does not have any adverse events (AEs), which would require IMP discontinuation.

Participants in this study will be required to make monthly visits to the study clinic and will be closely monitored over the course of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Male and female participants aged 4 to 17 years (inclusive) with a diagnosis of ADPKD as defined by the presence of family history and/or genetic criteria AND who have at least 10 renal cysts, each of which measure at least 0.5 cm, confirmed upon magnetic resonance imaging (MRI) inspection; participants under the age of 12 years must have at least 4 cysts that are at least 1 cm in size, confirmed by ultrasound.
* Weight ≥20 kg.
* Participants with estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73m^2 within 31 days prior to randomization (using the Schwartz formula, eGFR = 0.413 × height [cm]/serum creatinine milligrams per deciliter [mg/dL]).
* Independent in toileting.
* Ability to swallow a tablet.

Key Exclusion Criteria:

* Liver function tests including aspartate aminotransferase (AST), alanine aminotransferase (ALT) > 1.5 × the upper limit of normal (ULN).
* Nocturnal enuresis.
* Need for chronic diuretic use.
* Participants with advanced diabetes (e.g., glycosylated hemoglobin >7.5, and/or glycosuria by dipstick, significant proteinuria, retinopathy), evidence of additional significant renal disease(s) (i.e., currently active glomerular nephritides), renal cancer, single kidney, or recent (within 6 months of screening) renal surgery or acute kidney injury.
* Participants having disorders in thirst recognition or inability to access fluids.
* Participants with critical electrolyte imbalances, as determined by the investigator.
* Participants with, or at risk of, significant hypovolemia as determined by investigator.
* Participants with clinically significant anemia, as determined by investigator.
* Participants 12 years of age and older having contraindications to, or interference with MRI assessments (e.g., ferro-magnetic prostheses, aneurysm clips, severe claustrophobia).
* Participants with a history of taking a vasopressin agonist/antagonist.
* Participants taking medications or having concomitant illnesses likely to confound endpoint assessments, including taking approved (i.e., marketed) therapies for the purpose of affecting polycystic kidney disease (PKD) cysts such as tolvaptan, vasopressin antagonists, anti-sense ribonucleic acid (RNA) therapies, rapamycin, sirolimus, everolimus, or somatostatin analogs (i.e., octreotide, sandostatin).
* Participants who have had cyst reduction surgery within 6 weeks of the screening visit.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (17):
- Belgium (4):
  - Ghent, Oost-Vlaanderen
  - Leuven, Vlaams Brabant
  - Brussels
  - Montegnée
- Germany (6):
  - Cologne
  - Hamburg
  - Hanover
  - Heidelberg
  - Leipzig
  - Tübingen
- Italy (3):
  - Milan
  - Napoli
  - Pavia
- United Kingdom (4):
  - Birmingham
  - London
  - Manchester
  - Nottingham

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: https://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Shoaf SE, Sikes K. Tolvaptan pharmacokinetics and pharmacodynamics in adolescents with autosomal dominant polycystic kidney disease. Eur J Pediatr. 2025 Dec 18;185(1):26. doi: 10.1007/s00431-025-06689-2. PMID 41407907
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Mekahli D, Guay-Woodford LM, Cadnapaphornchai MA, Greenbaum LA, Litwin M, Seeman T, Dandurand A, Shi L, Sikes K, Shoaf SE, Schaefer F. Tolvaptan for Children and Adolescents with Autosomal Dominant Polycystic Kidney Disease: Randomized Controlled Trial. Clin J Am Soc Nephrol. 2023 Jan 1;18(1):36-46. doi: 10.2215/CJN.0000000000000022. PMID 36719158
- [Derived] Liu F, Feng C, Shen H, Fu H, Mao J. Tolvaptan in Pediatric Autosomal Dominant Polycystic Kidney Disease: From Here to Where? Kidney Dis (Basel). 2021 Sep;7(5):343-349. doi: 10.1159/000517186. Epub 2021 Jul 2. PMID 34604341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 18 sites in Belgium, Germany, Italy, and the United Kingdom from 23 September 2016 to 17 November 2021.
Pre-assignment Details: A total of 91 participants with autosomal dominant polycystic kidney disease (ADPKD) were randomized into 2 groups in a 1:1 ratio to receive tolvaptan or matching placebo.
Period: Phase A: Double-blind Period (12 Months)
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Started | 48 | 43 | 0 | 0
Dense Pharmacokinetic/Pharmacodynamic (PK/PD) Population (The Dense PK/PD Population included a subset of participants half on tolvaptan and half on placebo, in the 12 to 17 year old age group who had dense PK sampling after at least 1 month on IMP.) | 12 | 8 | 0 | 0
Completed | 44 | 40 | 0 | 0
Not Completed | 4 | 3 | 0 | 0
Not completed — Adverse Events | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 0 | 0
Period: Phase B: Open-label Period (24 Months)
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Started | 0 | 0 | 42 (2 Phase A: Tolvaptan completers did not enter Phase B.) | 39 (1 Phase A: Placebo completer did not enter Phase B.)
Completed | 0 | 0 | 36 | 33
Not Completed | 0 | 0 | 6 | 6
Not completed — Adverse Events | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 3
Not completed — Reason Not Specified | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Randomized Sample included all participants who were randomized in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Total
Number analyzed (Participants) | 48 | 43 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.9 (3.2) | 12.8 (2.8) | 12.9 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 27 | 20 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 47 | 42 | 89
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 46 | 42 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase A: Change From Baseline in Spot Urine Osmolality (Pre-morning Dose)
Description: Urine osmolality is a measure of urine concentration, measured by osmometer, which evaluates the freezing point depression of a solution and supplies results as milliosmoles per kilogram of water. Spot urine osmolality was determined for urine samples collected immediately prior to morning dosing for Day 1 (Baseline), and Week 1 for all participants. Sample was taken after the first morning's void and was provided as a mid-stream, clean catch sample. All participants were fasting.
Time Frame: Baseline, and Week 1 of Phase A
Population: The Full Analysis Set (FAS) included all participants who were randomized to a treatment group, received at least 1 dose of the investigational medicinal product (IMP), and had both a Phase A baseline and at least 1 postbaseline efficacy evaluation. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: milliosmoles per kilogram (mOsm/kg)
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 48 | 43
milliosmoles per kilogram (mOsm/kg)
  Baseline | 635 (252) | 646 (250)
  Change From Baseline at Week 1, Phase A: number analyzed (Participants) | 48 | 42
  Change From Baseline at Week 1, Phase A | -386 (284) | -93 (332)

2. Primary Outcome: Phase A: Change From Baseline in Specific Gravity (Pre-morning Dose)
Description: Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. Spot urine sample for determination of specific gravity was collected immediately prior to morning dosing for Day 1 (Baseline), and Week 1 for all participants. Sample was taken after the first morning's void and was provided as a mid-stream, clean catch sample. All participants were fasting.
Time Frame: Baseline, and Week 1 of Phase A
Population: The FAS included all participants who were randomized to a treatment group, received at least 1 dose of the IMP, and had both a Phase A baseline and at least 1 postbaseline efficacy evaluation. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 48 | 43
ratio
  Baseline | 1.017 (0.006) | 1.017 (0.006)
  Change From Baseline at Week 1, Phase A: number analyzed (Participants) | 48 | 41
  Change From Baseline at Week 1, Phase A | -0.009 (0.007) | -0.002 (0.008)

3. Secondary Outcome: Phase A: Percent Change From Phase A Baseline in Height-Adjusted Total Kidney Volume (htTKV) as Measured by Magnetic Resonance Imaging (MRI)
Description: htTKV is used in participants with autosomal dominant polycystic kidney disease to predict the onset of renal insufficiency.
Time Frame: Baseline, and Month 12 of Phase A
Population: The FAS included all participants who were randomized to a treatment group, received at least 1 dose of the IMP, and had both a Phase A baseline and at least 1 postbaseline efficacy evaluation. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 30 | 27
percent change | 2.28 (8.75) | 6.11 (7.48)

4. Secondary Outcome: Phase A and B: Mean 24-hour Fluid Balance Prior to Week 1
Description: Participants were instructed to record all fluid taken and all urine output for the 24-hour period.
Time Frame: Prior to Week 1 in Phase A and B
Population: The FAS for Phase A included all participants who were randomized to a treatment group, received at least 1 dose of the IMP, and had both a Phase A Baseline and at least 1 postbaseline efficacy evaluation. The FAS for Phase B included all participants who enrolled to Phase B, received at least 1 dose of the IMP, and had both a baseline and at least 1 postbaseline efficacy evaluation in Phase B. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 43 | 41 | 37 | 37
milliliter | 31 (1978) | 241 (867) | 138 (1382) | 207 (1355)

5. Secondary Outcome: Phase A: Change From Baseline in Renal Function (Estimated Glomerular Filtration Rate [eGFR] by Schwartz Formula) at Each Clinic Visit in Phase A
Description: Renal function was assessed by estimated eGFR calculated by the Schwartz formula (eGFR = 0.413 × height [cm] /serum creatinine mg/dL), expressed as mean change in eGFR at the specified time points. The units for the data reported are milliliter per minute per 1.73 meter square (mL/min/1.73 m^2). The baseline was the evaluation done at Week 1 in Phase A for this outcome measure.
Time Frame: Phase A Baseline, Months 1, 6, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 44 | 42
mL/min/1.73 m^2
  Baseline | 93.9 (18.7) | 102.1 (15.4)
  Change From Baseline at Month 1, Phase A: number analyzed (Participants) | 43 | 42
  Change From Baseline at Month 1, Phase A | 2.8 (10.7) | -1.9 (8.8)
  Change From Baseline at Month 6, Phase A: number analyzed (Participants) | 41 | 40
  Change From Baseline at Month 6, Phase A | 4.6 (10.1) | -2.5 (11.1)
  Change From Baseline at Month 12, Phase A: number analyzed (Participants) | 40 | 39
  Change From Baseline at Month 12, Phase A | 2.6 (10.7) | -3.2 (10.9)

6. Secondary Outcome: Phase B: Change From Phase B Baseline in Renal Function (eGFR by Schwartz Formula) at Each Clinic Visit in Phase B
Description: Renal function was assessed by estimated eGFR calculated by the Schwartz formula (eGFR = 0.413 × height [cm] /serum creatinine mg/dL), expressed as mean change in eGFR at the specified time points.
Time Frame: Phase B Baseline, Week 1, Months 1, 6, 12, 18, and 24
Population: The FAS for Phase B included all participants who enrolled to Phase B, received at least 1 dose of the IMP, and had both a baseline and at least 1 postbaseline efficacy evaluation in Phase B. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 42 | 39
mL/min/1.73 m^2
  Phase B Baseline | 97.0 (17.1) | 98.5 (14.1)
  Change From Phase B Baseline at Week 1, Phase B: number analyzed (Participants) | 40 | 37
  Change From Phase B Baseline at Week 1, Phase B | -1.7 (10.4) | -6.7 (8.0)
  Change From Phase B Baseline at Month 1, Phase B: number analyzed (Participants) | 41 | 38
  Change From Phase B Baseline at Month 1, Phase B | -0.9 (10.2) | -4.8 (9.0)
  Change From Phase B Baseline at Month 6, Phase B: number analyzed (Participants) | 38 | 33
  Change From Phase B Baseline at Month 6, Phase B | -4.2 (9.6) | -6.4 (7.9)
  Change From Phase B Baseline at Month 12, Phase B: number analyzed (Participants) | 36 | 36
  Change From Phase B Baseline at Month 12, Phase B | -5.6 (11.1) | -7.2 (9.3)
  Change From Phase B Baseline at Month 18, Phase B: number analyzed (Participants) | 29 | 27
  Change From Phase B Baseline at Month 18, Phase B | -3.5 (9.8) | -9.0 (10.9)
  Change From Phase B Baseline at Month 24, Phase B: number analyzed (Participants) | 34 | 31
  Change From Phase B Baseline at Month 24, Phase B | -5.2 (9.4) | -10.3 (11.0)

7. Secondary Outcome: Phase B: Percent Change From Phase B Baseline in htTKV as Measured by MRI at Month 12 and Month 24
Description: as for outcome 3
Time Frame: Phase B Baseline, Months 12 and 24
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 26 | 23
percent change
  Percent Change From Phase B Baseline at Month 12, Phase B | 7.68 (9.67) | 3.09 (8.97)
  Percent Change From Phase B Baseline at Month 24 Phase B: number analyzed (Participants) | 24 | 21
  Percent Change From Phase B Baseline at Month 24 Phase B | 13.55 (12.88) | 7.35 (9.57)

8. Secondary Outcome: Phase A: 24-hour Urine Volume
Description: Urine volume refers to the quantity of urine produced per unit of time.
Time Frame: 24 hours post dose after Month 1 on study medication in Phase A
Population: The Dense Pharmacokinetic/Pharmacodynamic (PK/PD) Population included a subset of participants half on tolvaptan and half on placebo, in the 12 to 17 year old age group who had dense PK sampling after at least 1 month on IMP. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: milliliter per 24 hours post dose
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 12 | 8
milliliter per 24 hours post dose | 7171 (2810) | 2529 (2164)

9. Secondary Outcome: Phase A: 24-hour Fluid Intake
Description: Daily fluid intake (total water) is defined as the amount of water consumed from foods, plain drinking water, and other beverages.
Time Frame: 24 hours post dose after Month 1 on study medication in Phase A
Population: The Dense PK/PD Population included a subset of participants half on tolvaptan and half on placebo, in the 12 to 17 year old age group who had dense PK sampling after at least 1 month on IMP. Overall number analyzed are the number of participants with data available for analyses.
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 11 | 5
milliliter | 7486 (2350) | 3156 (1775)

10. Secondary Outcome: Phase A: 24-hour Fluid Balance
Description: Fluid balance is a term used to describe the balance of the input and output of fluids in the body to allow metabolic processes to function correctly.
Time Frame: 24 hours post dose after Month 1 on study medication in Phase A
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: milliliter
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 11 | 5
milliliter | 53 (1894) | 230 (1254)

11. Secondary Outcome: Phase A: 24-hour Sodium Clearance
Description: Data was categorized and reported based on the total daily dose for the given time point of 0-24 hours.
Time Frame: 24 hours post dose after Month 1 on study medication in Phase A
Population: The Dense PK/PD Population included a subset of participants half on tolvaptan and half on placebo, in the 12 to 17 year old age group who had dense PK sampling after at least 1 month on IMP. Overall number analyzed are the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Mean (Standard Deviation); unit: milliliter per minute (mL/min)
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 10 | 7
milliliter per minute (mL/min)
  Total Daily Dose: 37.5 mg: number analyzed (Participants) | 3 | 0
  Total Daily Dose: 37.5 mg | 0.8 (0.3) |
  Total Daily Dose: 45 mg: number analyzed (Participants) | 3 | 0
  Total Daily Dose: 45 mg | 0.7 (0.3) |
  Total Daily Dose: 60 mg: number analyzed (Participants) | 4 | 0
  Total Daily Dose: 60 mg | 0.9 (0.3) |
  Total Daily Dose: Placebo: number analyzed (Participants) | 0 | 7
  Total Daily Dose: Placebo |  | 0.7 (0.5)

12. Secondary Outcome: Phase A: 24-hour Creatinine Clearance
Description: Creatinine is produced from the metabolism of protein, when muscles burn energy. Most creatinine is filtered out of the blood by the kidneys and excreted in urine. The creatinine clearance value is determined by measuring the concentration of endogenous creatinine (that which is produced by the body) in both plasma and urine. Data was categorized and reported based on the total daily dose for the given time point of 0-24 hours.
Time Frame: 24 hours post dose after Month 1 on study medication in Phase A
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 11 | 8
mL/min
  Total Daily Dose: 22.5 mg: number analyzed (Participants) | 1 | 0
  Total Daily Dose: 22.5 mg | 124.6 (NA) — The standard deviation was not estimable due to lower number of participants with event. |
  Total Daily Dose: 37.5 mg: number analyzed (Participants) | 3 | 0
  Total Daily Dose: 37.5 mg | 148.5 (23.4) |
  Total Daily Dose: 45 mg: number analyzed (Participants) | 3 | 0
  Total Daily Dose: 45 mg | 95.0 (10.1) |
  Total Daily Dose: 60 mg: number analyzed (Participants) | 4 | 0
  Total Daily Dose: 60 mg | 123.7 (23.2) |
  Total Daily Dose: Placebo: number analyzed (Participants) | 0 | 8
  Total Daily Dose: Placebo |  | 105.1 (51.7)

13. Secondary Outcome: Phase A: 24-hour Free Water Clearance
Description: Data was categorized and reported based on the total daily dose for the given time point of 0-24 hours.
Time Frame: 24 hours post dose after Month 1 on study medication in Phase A
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 11 | 8
mL/min
  Total Daily Dose: 37.5 mg: number analyzed (Participants) | 3 | 0
  Total Daily Dose: 37.5 mg | 2.3 (0.9) |
  Total Daily Dose: 45 mg: number analyzed (Participants) | 3 | 0
  Total Daily Dose: 45 mg | 2.6 (0.9) |
  Total Daily Dose: 60 mg: number analyzed (Participants) | 5 | 0
  Total Daily Dose: 60 mg | 3.0 (1.2) |
  Total Daily Dose: Placebo: number analyzed (Participants) | 0 | 8
  Total Daily Dose: Placebo |  | 0.1 (1.2)

14. Secondary Outcome: Phase A: Percentage of Each Tanner Stage by Gender and Age Compared to Normative Populations
Description: Tanner stages is a scale that defines physical measurements of development based on external primary and secondary sex characteristics. It was used in this study to assess pubertal development with values ranging from Stage 1 (pre-pubertal characteristics) to Stage 5 (adult or mature characteristics). Only those categories with at least one participant with event are reported.
Time Frame: At Baseline, Months 6 and 12 of Phase A
Population: The Phase A Safety Set included all participants who were randomized and received at least 1 dose of IMP in Phase A.
Measure: Number; unit: percentage of participants
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 48 | 43
percentage of participants
  Female (>=4 to <12 Years): Baseline- Stage 1 | 6.3 | 11.6
  Female (>=4 to <12 Years): Baseline- Stage 3 | 0.0 | 2.3
  Female (>=4 to <12 Years): Month 6, Phase A- Stage 1 | 6.3 | 9.3
  Female (>=4 to <12 Years): Month 6, Phase A- Stage 2 | 0.0 | 2.3
  Female (>=4 to <12 Years): Month 6, Phase A- Stage 4 | 0.0 | 2.3
  Female (>=4 to <12 Years): Month 12, Phase A- Stage 1 | 4.2 | 7.0
  Female (>=4 to <12 Years): Month 12, Phase A- Stage 2 | 0.0 | 2.3
  Female (>=4 to <12 Years): Month 12, Phase A- Stage 4 | 0.0 | 2.3
  Male (>=4 to <12 Years): Baseline- Stage 1 | 16.7 | 4.7
  Male (>=4 to <12 Years): Baseline- Stage 2 | 0.0 | 4.7
  Male (>=4 to <12 Years): Baseline- Stage 3 | 2.1 | 0.0
  Male (>=4 to <12 Years): Month 6, Phase A- Stage 1 | 16.7 | 7.0
  Male (>=4 to <12 Years): Month 6, Phase A- Stage 2 | 2.1 | 0.0
  Male (>=4 to <12 Years): Month 6, Phase A- Stage 3 | 2.1 | 4.7
  Male (>=4 to <12 Years): Month 12, Phase A- Stage 1 | 14.6 | 4.7
  Male (>=4 to <12 Years): Month 12, Phase A- Stage 2 | 4.2 | 2.3
  Male (>=4 to <12 Years): Month 12, Phase A- Stage 3 | 0.0 | 4.7
  Male (>=4 to <12 Years): Month 12, Phase A- Stage 4 | 2.1 | 0.0
  Female (>=12 to <15 Years): Baseline- Stage 1 | 2.1 | 0.0
  Female (>=12 to <15 Years): Baseline- Stage 2 | 0.0 | 4.7
  Female (>=12 to <15 Years): Baseline- Stage 3 | 2.1 | 2.3
  Female (>=12 to <15 Years): Baseline- Stage 4 | 4.2 | 0.0
  Female (>=12 to <15 Years): Baseline- Stage 5 | 10.4 | 7.0
  Female (>=12 to <15 Years): Month 6, Phase A- Stage 2 | 0.0 | 2.3
  Female (>=12 to <15 Years): Month 6, Phase A- Stage 3 | 0.0 | 2.3
  Female (>=12 to <15 Years): Month 6, Phase A- Stage 4 | 2.1 | 0.0
  Female (>=12 to <15 Years): Month 6, Phase A- Stage 5 | 12.5 | 7.0
  Female (>=12 to <15 Years): Month 12, Phase A- Stage 2 | 0.0 | 2.3
  Female (>=12 to <15 Years): Month 12, Phase A- Stage 3 | 0.0 | 2.3
  Female (>=12 to <15 Years): Month 12, Phase A- Stage 4 | 0.0 | 4.7
  Female (>=12 to <15 Years): Month 12, Phase A- Stage 5 | 14.6 | 9.3
  Male (>=12 to <15 Years): Baseline- Stage 2 | 6.3 | 4.7
  Male (>=12 to <15 Years): Baseline- Stage 3 | 4.2 | 4.7
  Male (>=12 to <15 Years): Baseline- Stage 4 | 2.1 | 4.7
  Male (>=12 to <15 Years): Baseline- Stage 5 | 2.1 | 2.3
  Male (>=12 to <15 Years): Month 6, Phase A- Stage 2 | 4.2 | 2.3
  Male (>=12 to <15 Years): Month 6, Phase A- Stage 3 | 4.2 | 2.3
  Male (>=12 to <15 Years): Month 6, Phase A- Stage 4 | 4.2 | 4.7
  Male (>=12 to <15 Years): Month 6, Phase A- Stage 5 | 2.1 | 2.3
  Male (>=12 to <15 Years): Month 12, Phase A- Stage 2 | 0.0 | 2.3
  Male (>=12 to <15 Years): Month 12, Phase A- Stage 3 | 2.1 | 0.0
  Male (>=12 to <15 Years): Month 12, Phase A- Stage 4 | 8.3 | 7.0
  Male (>=12 to <15 Years): Month 12, Phase A- Stage 5 | 4.2 | 2.3
  Male (>=12 to <15 Years): End of Treatment- Stage 5 | 2.1 | 2.3
  Female (>=15 to <18 Years): Baseline- Stage 4 | 2.1 | 0.0
  Female (>=15 to <18 Years): Baseline- Stage 5 | 12.5 | 18.6
  Female (>=15 to <18 Years): Month 6, Phase A- Stage 4 | 2.1 | 0.0
  Female (>=15 to <18 Years): Month 6, Phase A- Stage 5 | 12.5 | 16.3
  Female (>=15 to <18 Years): Month 12, Phase A- Stage 4 | 2.1 | 0.0
  Female (>=15 to <18 Years): Month 12, Phase A- Stage 5 | 14.6 | 16.3
  Female (>=15 to <18 Years): End of Treatment- Stage 5 | 0.0 | 2.3
  Male (>=15 to <18 Years): Baseline- Stage 4 | 2.1 | 4.7
  Male (>=15 to <18 Years): Baseline- Stage 5 | 16.7 | 14.0
  Male (>=15 to <18 Years): Month 6, Phase A- Stage 4 | 2.1 | 2.3
  Male (>=15 to <18 Years): Month 6, Phase A- Stage 5 | 14.6 | 16.3
  Male (>=15 to <18 Years): Month 12, Phase A- Stage 4 | 2.1 | 0.0
  Male (>=15 to <18 Years): Month 12, Phase A- Stage 5 | 14.6 | 18.6
  Male (>=15 to <18 Years): End of Treatment- Stage 5 | 2.1 | 0.0

15. Secondary Outcome: Phase B: Percentage of Each Tanner Stage by Gender and Age Compared to Normative Populations
Description: as for outcome 14
Time Frame: At Baseline, Months 6, 12, 18, and 24 of Phase B
Population: The Phase B Safety Set included all participants who were enrolled in Phase B and received at least 1 dose of IMP in Phase B.
Measure: Number; unit: percentage of participants
Arm/Group | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 42 | 39
percentage of participants
  Female (>=4 to <12 Years): Phase B Baseline- Stage 1 | 7.1 | 10.3
  Female (>=4 to <12 Years): Phase B Baseline- Stage 2 | 0.0 | 2.6
  Female (>=4 to <12 Years): Phase B Baseline- Stage 4 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 6, Phase B- Stage 1 | 4.8 | 7.7
  Female (>=4 to <12 Years): Month 6, Phase B- Stage 2 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 6, Phase B- Stage 4 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 12, Phase B- Stage 1 | 4.8 | 7.7
  Female (>=4 to <12 Years): Month 12, Phase B- Stage 2 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 12, Phase B- Stage 3 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 12, Phase B- Stage 4 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 18, Phase B- Stage 1 | 4.8 | 2.6
  Female (>=4 to <12 Years): Month 18, Phase B- Stage 2 | 0.0 | 7.7
  Female (>=4 to <12 Years): Month 18, Phase B- Stage 4 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 24, Phase B- Stage 1 | 2.4 | 2.6
  Female (>=4 to <12 Years): Month 24, Phase B- Stage 2 | 2.4 | 5.1
  Female (>=4 to <12 Years): Month 24, Phase B- Stage 3 | 0.0 | 2.6
  Female (>=4 to <12 Years): Month 24, Phase B- Stage 4 | 0.0 | 2.6
  Male (>=4 to <12 Years): Phase B Baseline- Stage 1 | 11.9 | 5.1
  Male (>=4 to <12 Years): Phase B Baseline- Stage 2 | 4.8 | 2.6
  Male (>=4 to <12 Years): Phase B Baseline- Stage 3 | 0.0 | 5.1
  Male (>=4 to <12 Years): Phase B Baseline- Stage 4 | 2.4 | 0.0
  Male (>=4 to <12 Years): Month 6, Phase B- Stage 1 | 9.5 | 2.6
  Male (>=4 to <12 Years): Month 6, Phase B- Stage 2 | 2.4 | 2.6
  Male (>=4 to <12 Years): Month 6, Phase B- Stage 3 | 2.4 | 2.6
  Male (>=4 to <12 Years): Month 6, Phase B- Stage 4 | 2.4 | 2.6
  Male (>=4 to <12 Years): Month 12, Phase B- Stage 1 | 9.5 | 2.6
  Male (>=4 to <12 Years): Month 12, Phase B- Stage 2 | 2.4 | 0.0
  Male (>=4 to <12 Years): Month 12, Phase B- Stage 3 | 2.4 | 5.1
  Male (>=4 to <12 Years): Month 12, Phase B- Stage 4 | 2.4 | 2.6
  Male (>=4 to <12 Years): Month 18, Phase B- Stage 1 | 4.8 | 2.6
  Male (>=4 to <12 Years): Month 18, Phase B- Stage 2 | 2.4 | 0.0
  Male (>=4 to <12 Years): Month 18, Phase B- Stage 3 | 0.0 | 5.1
  Male (>=4 to <12 Years): Month 18, Phase B- Stage 4 | 4.8 | 0.0
  Male (>=4 to <12 Years): Month 18, Phase B- Stage 5 | 0.0 | 2.6
  Male (>=4 to <12 Years): Month 24, Phase B- Stage 1 | 4.8 | 0.0
  Male (>=4 to <12 Years): Month 24, Phase B- Stage 2 | 4.8 | 0.0
  Male (>=4 to <12 Years): Month 24, Phase B- Stage 3 | 2.4 | 5.1
  Male (>=4 to <12 Years): Month 24, Phase B- Stage 4 | 2.4 | 0.0
  Male (>=4 to <12 Years): Month 24, Phase B- Stage 5 | 2.4 | 2.6
  Female (>=12 to <15 Years): Phase B Baseline- Stage 2 | 0.0 | 2.6
  Female (>=12 to <15 Years): Phase B Baseline- Stage 3 | 0.0 | 2.6
  Female (>=12 to <15 Years): Phase B Baseline- Stage 4 | 0.0 | 5.1
  Female (>=12 to <15 Years): Phase B Baseline- Stage 5 | 16.7 | 10.3
  Female (>=12 to <15 Years): Month 6, Phase B- Stage 3 | 0.0 | 5.1
  Female (>=12 to <15 Years): Month 6, Phase B- Stage 4 | 0.0 | 5.1
  Female (>=12 to <15 Years): Month 6, Phase B-Stage 5 | 16.7 | 10.3
  Female (>=12 to <15 Years): Month 12, Phase B- Stage 4 | 0.0 | 5.1
  Female (>=12 to <15 Years): Month 12, Phase B- Stage 5 | 14.3 | 10.3
  Female (>=12 to <15 Years): Month 18, Phase B- Stage 4 | 0.0 | 2.6
  Female (>=12 to <15 Years): Month 18, Phase B- Stage 5 | 11.9 | 10.3
  Female (>=12 to <15 Years): Month 24, Phase B- Stage 4 | 0.0 | 5.1
  Female (>=12 to <15 Years): Month 24, Phase B- Stage 5 | 9.5 | 10.3
  Female (>=12 to <15 Years): End of Treatment, Phase B- Stage 4 | 0.0 | 2.6
  Female (>=12 to <15 Years): End of Treatment, Phase B- Stage 5 | 7.1 | 2.6
  Male (>=12 to <15 Years): Phase B Baseline- Stage 2 | 0.0 | 2.6
  Male (>=12 to <15 Years): Phase B Baseline- Stage 3 | 2.4 | 0.0
  Male (>=12 to <15 Years): Phase B Baseline- Stage 4 | 9.5 | 7.7
  Male (>=12 to <15 Years): Phase B Baseline- Stage 5 | 4.8 | 2.6
  Male (>=12 to <15 Years): Month 6, Phase B- Stage 2 | 0.0 | 2.6
  Male (>=12 to <15 Years): Month 6, Phase B- Stage 3 | 2.4 | 0.0
  Male (>=12 to <15 Years): Month 6, Phase B- Stage 4 | 4.8 | 5.1
  Male (>=12 to <15 Years): Month 6, Phase B- Stage 5 | 4.8 | 2.6
  Male (>=12 to <15 Years): Month 12, Phase B- Stage 2 | 0.0 | 2.6
  Male (>=12 to <15 Years): Month 12, Phase B- Stage 4 | 7.1 | 5.1
  Male (>=12 to <15 Years): Month 12, Phase B- Stage 5 | 7.1 | 5.1
  Male (>=12 to <15 Years): Month 18, Phase B- Stage 2 | 0.0 | 2.6
  Male (>=12 to <15 Years): Month 18, Phase B- Stage 4 | 4.8 | 0.0
  Male (>=12 to <15 Years): Month 18, Phase B- Stage 5 | 9.5 | 7.7
  Male (>=12 to <15 Years): Month 24, Phase B- Stage 2 | 0.0 | 2.6
  Male (>=12 to <15 Years): Month 24, Phase B- Stage 4 | 4.8 | 0.0
  Male (>=12 to <15 Years): Month 24, Phase B- Stage 5 | 9.5 | 10.3
  Male (>=12 to <15 Years): End of Treatment, Phase B- Stage 5 | 0.0 | 2.6
  Female (>=15 to <18 Years): Phase B Baseline- Stage 4 | 2.4 | 0.0
  Female (>=15 to <18 Years): Phase B Baseline- Stage 5 | 16.7 | 15.4
  Female (>=15 to <18 Years): Month 6, Phase B- Stage 4 | 2.4 | 0.0
  Female (>=15 to <18 Years): Month 6, Phase B- Stage 5 | 16.7 | 12.8
  Female (>=15 to <18 Years): Month 12, Phase B- Stage 4 | 2.4 | 0.0
  Female (>=15 to <18 Years): Month 12, Phase B- Stage 5 | 16.7 | 12.8
  Female (>=15 to <18 Years): Month 18, Phase B- Stage 4 | 2.4 | 0.0
  Female (>=15 to <18 Years): Month 18, Phase B- Stage 5 | 16.7 | 12.8
  Female (>=15 to <18 Years): Month 24, Phase B- Stage 4 | 2.4 | 0.0
  Female (>=15 to <18 Years): Month 24, Phase B- Stage 5 | 16.7 | 12.8
  Female (>=15 to <18 Years): End of Treatment, Phase B- Stage 5 | 0.0 | 5.1
  Male (>=15 to <18 Years): Phase B Baseline- Stage 4 | 2.4 | 0.0
  Male (>=15 to <18 Years): Phase B Baseline- Stage 5 | 16.7 | 20.5
  Male (>=15 to <18 Years): Month 6, Phase B- Stage 5 | 19.0 | 17.9
  Male (>=15 to <18 Years): Month 12, Phase B- Stage 5 | 16.7 | 17.9
  Male (>=15 to <18 Years): Month 18, Phase B- Stage 5 | 16.7 | 15.4
  Male (>=15 to <18 Years): Month 24, Phase B- Stage 5 | 16.7 | 12.8
  Male (>=15 to <18 Years): End of Treatment, Phase B- Stage 5 | 4.8 | 7.7

16. Secondary Outcome: Phase A: Change From Baseline in Growth Percentile by Gender and Age
Description: The growth percentile was based on the assessment of height and weight.
Time Frame: At Baseline, Months 6 and 12 of Phase A
Population: The Phase A Safety Set included all participants who were randomized and received at least 1 dose of IMP in Phase A. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: growth percentile
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 48 | 43
growth percentile
  Female Participants with Age >=15 to <18 Years - Baseline, Phase A: number analyzed (Participants) | 9 | 8
  Female Participants with Age >=15 to <18 Years - Baseline, Phase A | 62 (28) | 60 (34)
  Change From Baseline in Female Participants with Age >=15 to <18 Years - Month 6, Phase A: number analyzed (Participants) | 9 | 6
  Change From Baseline in Female Participants with Age >=15 to <18 Years - Month 6, Phase A | 2 (18) | -2 (12)
  Change From Baseline in Female Participants with Age >=15 to <18 Years - Month 12, Phase A: number analyzed (Participants) | 9 | 7
  Change From Baseline in Female Participants with Age >=15 to <18 Years - Month 12, Phase A | 7 (10) | -5 (11)
  Male Participants with Age >=15 to <18 Years - Baseline, Phase A: number analyzed (Participants) | 9 | 8
  Male Participants with Age >=15 to <18 Years - Baseline, Phase A | 56 (29) | 73 (18)
  Change From Baseline in Male Participants with Age >=15 to <18 Years - Month 6, Phase A: number analyzed (Participants) | 8 | 8
  Change From Baseline in Male Participants with Age >=15 to <18 Years - Month 6, Phase A | 12 (16) | -1 (30)
  Change From Baseline in Male Participants with Age >=15 to <18 Years - Month 12, Phase A: number analyzed (Participants) | 8 | 8
  Change From Baseline in Male Participants with Age >=15 to <18 Years - Month 12, Phase A | 2 (37) | -3 (25)
  Female Participants with Age >=12 to <15 Years - Baseline, Phase A: number analyzed (Participants) | 9 | 8
  Female Participants with Age >=12 to <15 Years - Baseline, Phase A | 71 (20) | 72 (29)
  Change From Baseline in Female Participants with Age >=12 to <15 Years - Month 6, Phase A: number analyzed (Participants) | 7 | 8
  Change From Baseline in Female Participants with Age >=12 to <15 Years - Month 6, Phase A | -2 (12) | -20 (21)
  Change From Baseline in Female Participants with Age >=12 to <15 Years - Month 12, Phase A: number analyzed (Participants) | 7 | 8
  Change From Baseline in Female Participants with Age >=12 to <15 Years - Month 12, Phase A | -11 (9) | -18 (27)
  Male Participants with Age >=12 to <15 Years - Baseline, Phase A: number analyzed (Participants) | 8 | 7
  Male Participants with Age >=12 to <15 Years - Baseline, Phase A | 70 (21) | 76 (24)
  Change From Baseline in Male Participants with Age >=12 to <15 Years - Month 6, Phase A: number analyzed (Participants) | 7 | 7
  Change From Baseline in Male Participants with Age >=12 to <15 Years - Month 6, Phase A | -7 (13) | -13 (38)
  Change From Baseline in Male Participants with Age >=12 to <15 Years - Month 12, Phase A: number analyzed (Participants) | 7 | 5
  Change From Baseline in Male Participants with Age >=12 to <15 Years - Month 12, Phase A | 0 (20) | 8 (17)
  Female Participants with Age 4 to <=11 Years - Baseline, Phase A: number analyzed (Participants) | 3 | 7
  Female Participants with Age 4 to <=11 Years - Baseline, Phase A | 71 (25) | 57 (14)
  Change From Baseline in Female Participants with Age 4 to <=11 Years - Month 6, Phase A: number analyzed (Participants) | 3 | 7
  Change From Baseline in Female Participants with Age 4 to <=11 Years - Month 6, Phase A | -1 (3) | 4 (16)
  Change From Baseline in Female Participants with Age 4 to <=11 Years - Month 12, Phase A: number analyzed (Participants) | 3 | 7
  Change From Baseline in Female Participants with Age 4 to <=11 Years - Month 12, Phase A | 7 (15) | 2 (18)
  Male Participants with Age 4 to <=11 Years - Baseline, Phase A: number analyzed (Participants) | 10 | 5
  Male Participants with Age 4 to <=11 Years - Baseline, Phase A | 57 (31) | 63 (19)
  Change From Baseline in Male Participants with Age 4 to <=11 Years - Month 6, Phase A: number analyzed (Participants) | 10 | 5
  Change From Baseline in Male Participants with Age 4 to <=11 Years - Month 6, Phase A | 4 (16) | 0 (0)
  Change From Baseline in Male Participants with Age 4 to <=11 Years - Month 12, Phase A: number analyzed (Participants) | 10 | 5
  Change From Baseline in Male Participants with Age 4 to <=11 Years - Month 12, Phase A | 1 (3) | 1 (4)

17. Secondary Outcome: Phase B: Change From Baseline in Growth Percentile by Gender and Age
Description: The growth percentile was based on the assessment of height and weight.
Time Frame: At Baseline, Months 6, 12, 18, and 24 of Phase B
Population: The Phase B Safety Set included all participants who were enrolled in Phase B and received at least 1 dose of IMP in Phase B. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: growth percentile
Arm/Group | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 42 | 39
growth percentile
  Female Participants with Age >=15 to <18 Years - Phase B Baseline: number analyzed (Participants) | 9 | 6
  Female Participants with Age >=15 to <18 Years - Phase B Baseline | 69 (32) | 46 (28)
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 6, Phase B: number analyzed (Participants) | 7 | 5
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 6, Phase B | -7 (17) | 12 (21)
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 12, Phase B: number analyzed (Participants) | 8 | 5
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 12, Phase B | 0 (7) | 20 (18)
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 18, Phase B: number analyzed (Participants) | 6 | 3
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 18, Phase B | -2 (2) | 10 (9)
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 24, Phase B: number analyzed (Participants) | 8 | 5
  Change From Baseline Female Participants with Age >=15 to <18 Years - Month 24, Phase B | 6 (16) | 16 (20)
  Male Participants with Age >=15 to <18 Years - Phase B Baseline: number analyzed (Participants) | 8 | 8
  Male Participants with Age >=15 to <18 Years - Phase B Baseline | 60 (34) | 69 (18)
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 6, Phase B: number analyzed (Participants) | 8 | 7
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 6, Phase B | -13 (53) | 1 (2)
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 12, Phase B: number analyzed (Participants) | 6 | 6
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 12, Phase B | -8 (47) | 8 (11)
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 18, Phase B: number analyzed (Participants) | 5 | 6
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 18, Phase B | 16 (65) | -4 (25)
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 24, Phase B: number analyzed (Participants) | 6 | 5
  Change From Baseline Male Participants with Age >=15 to <18 Years - Month 24, Phase B | -2 (50) | -11 (25)
  Female Participants with Age >=12 to <15 Years - Phase B Baseline: number analyzed (Participants) | 7 | 8
  Female Participants with Age >=12 to <15 Years - Phase B Baseline | 62 (24) | 54 (34)
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 6, Phase B: number analyzed (Participants) | 7 | 8
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 6, Phase B | 3 (6) | 13 (18)
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 12, Phase B: number analyzed (Participants) | 6 | 8
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 12, Phase B | 12 (20) | 12 (23)
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 18, Phase B: number analyzed (Participants) | 5 | 5
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 18, Phase B | 5 (9) | 10 (22)
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 24, Phase B: number analyzed (Participants) | 4 | 7
  Change From Baseline Female Participants with Age >=12 to <15 Years - Month 24, Phase B | 1 (3) | 13 (18)
  Male Participants with Age >=12 to <15 Years - Phase B Baseline: number analyzed (Participants) | 7 | 5
  Male Participants with Age >=12 to <15 Years - Phase B Baseline | 67 (26) | 77 (23)
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 6, Phase B: number analyzed (Participants) | 5 | 5
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 6, Phase B | 1 (10) | -15 (38)
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 12, Phase B: number analyzed (Participants) | 7 | 5
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 12, Phase B | 4 (16) | -23 (37)
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 18, Phase B: number analyzed (Participants) | 5 | 4
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 18, Phase B | -4 (14) | -22 (40)
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 24, Phase B: number analyzed (Participants) | 6 | 5
  Change From Baseline Male Participants with Age >=12 to <15 Years - Month 24, Phase B | -8 (15) | -18 (36)
  Female Participants with Age 4 to <=11 Years - Phase B Baseline: number analyzed (Participants) | 3 | 7
  Female Participants with Age 4 to <=11 Years - Phase B Baseline | 78 (19) | 59 (22)
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 6, Phase B: number analyzed (Participants) | 3 | 6
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 6, Phase B | -2 (2) | 2 (12)
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 12, Phase B: number analyzed (Participants) | 3 | 7
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 12, Phase B | 5 (8) | 1 (12)
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 18, Phase B: number analyzed (Participants) | 3 | 7
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 18, Phase B | -5 (6) | 2 (23)
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 24, Phase B: number analyzed (Participants) | 3 | 7
  Change From Baseline Female Participants with Age 4 to <=11 Years - Month 24, Phase B | -4 (5) | 10 (21)
  Male Participants with Age 4 to <=11 Years - Phase B Baseline: number analyzed (Participants) | 8 | 5
  Male Participants with Age 4 to <=11 Years - Phase B Baseline | 65 (30) | 64 (21)
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 6, Phase B: number analyzed (Participants) | 8 | 4
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 6, Phase B | 0 (13) | 1 (2)
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 12, Phase B: number analyzed (Participants) | 8 | 5
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 12, Phase B | 3 (20) | 4 (8)
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 18, Phase B: number analyzed (Participants) | 5 | 4
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 18, Phase B | -4 (12) | 2 (9)
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 24, Phase B: number analyzed (Participants) | 7 | 4
  Change From Baseline Male Participants with Age 4 to <=11 Years - Month 24, Phase B | 0 (18) | 21 (23)

18. Secondary Outcome: Phase A: Change From Baseline in Creatinine Value
Description: Phase A Baseline is the last pre-dose evaluation. The Last Visit is the last available post-baseline evaluation including early term. As prespecified in the protocol, data for safety is reported by the treatment group (Phase A: Tolvaptan and Phase A: Placebo)
Time Frame: Baseline, Week 1, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, Follow Up Day 7, End of Treatment, and Last Visit
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo
Number analyzed (Participants) | 48 | 43
milligrams per deciliter (mg/dL)
  Baseline | 0.70 (0.16) | 0.67 (0.12)
  Change From Baseline at Week 1: number analyzed (Participants) | 47 | 42
  Change From Baseline at Week 1 | 0.04 (0.09) | -0.01 (0.06)
  Change From Baseline at Month 1 | 0.01 (0.08) | 0.01 (0.06)
  Change From Baseline at Month 2: number analyzed (Participants) | 44 | 42
  Change From Baseline at Month 2 | 0.01 (0.09) | 0.00 (0.07)
  Change From Baseline at Month 3: number analyzed (Participants) | 45 | 43
  Change From Baseline at Month 3 | 0.00 (0.11) | 0.01 (0.06)
  Change From Baseline at Month 4: number analyzed (Participants) | 45 | 40
  Change From Baseline at Month 4 | 0.00 (0.09) | -0.01 (0.07)
  Change From Baseline at Month 5: number analyzed (Participants) | 45 | 39
  Change From Baseline at Month 5 | 0.01 (0.09) | 0.01 (0.06)
  Change From Baseline at Month 6: number analyzed (Participants) | 44 | 41
  Change From Baseline at Month 6 | 0.01 (0.10) | 0.02 (0.07)
  Change From Baseline at Month 7: number analyzed (Participants) | 44 | 39
  Change From Baseline at Month 7 | 0.01 (0.10) | 0.02 (0.06)
  Change From Baseline at Month 8: number analyzed (Participants) | 43 | 39
  Change From Baseline at Month 8 | 0.01 (0.11) | 0.02 (0.07)
  Change From Baseline at Month 9: number analyzed (Participants) | 44 | 39
  Change From Baseline at Month 9 | 0.04 (0.11) | 0.01 (0.07)
  Change From Baseline at Month 10: number analyzed (Participants) | 40 | 34
  Change From Baseline at Month 10 | 0.01 (0.10) | 0.03 (0.07)
  Change From Baseline at Month 11: number analyzed (Participants) | 41 | 38
  Change From Baseline at Month 11 | 0.02 (0.11) | 0.04 (0.08)
  Change From Baseline at Month 12: number analyzed (Participants) | 43 | 40
  Change From Baseline at Month 12 | 0.02 (0.09) | 0.02 (0.06)
  Change From Baseline at Follow Up Day 7: number analyzed (Participants) | 1 | 1
  Change From Baseline at Follow Up Day 7 | 0.09 (NA) — The standard deviation was not estimable due to lower number of participants with event. | -0.02 (NA) — The standard deviation was not estimable due to lower number of participants with event.
  Change From Baseline at End of Treatment: number analyzed (Participants) | 2 | 3
  Change From Baseline at End of Treatment | 0.03 (0.10) | 0.03 (0.04)
  Change From Baseline at Last Visit | 0.03 (0.09) | 0.02 (0.06)

19. Secondary Outcome: Phase B: Change From Baseline in Creatinine Value
Description: Phase B Baseline is the last evaluation prior to the first dose in Phase B. The Last Visit is the last available post-baseline evaluation including early term. As prespecified in the protocol, data for safety is reported by the treatment group (Phase B: Prior Tolvaptan and Phase B: Prior Placebo).
Time Frame: Baseline, Week 1, Months 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, Follow Up Day 7, End of Treatment, and Last Visit
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 42 | 39
mg/dL
  Baseline | 0.73 (0.17) | 0.69 (0.13)
  Change From Baseline at Week 1: number analyzed (Participants) | 42 | 38
  Change From Baseline at Week 1 | 0.01 (0.06) | 0.04 (0.06)
  Change From Baseline at Month 1: number analyzed (Participants) | 41 | 38
  Change From Baseline at Month 1 | 0.01 (0.07) | 0.04 (0.06)
  Change From Baseline at Month 2: number analyzed (Participants) | 41 | 37
  Change From Baseline at Month 2 | 0.02 (0.07) | 0.04 (0.07)
  Change From Baseline at Month 3: number analyzed (Participants) | 41 | 37
  Change From Baseline at Month 3 | 0.02 (0.07) | 0.04 (0.07)
  Change From Baseline at Month 4: number analyzed (Participants) | 40 | 36
  Change From Baseline at Month 4 | 0.04 (0.06) | 0.05 (0.07)
  Change From Baseline at Month 5: number analyzed (Participants) | 38 | 30
  Change From Baseline at Month 5 | 0.03 (0.06) | 0.07 (0.07)
  Change From Baseline at Month 6: number analyzed (Participants) | 38 | 33
  Change From Baseline at Month 6 | 0.03 (0.07) | 0.06 (0.07)
  Change From Baseline at Month 7: number analyzed (Participants) | 38 | 32
  Change From Baseline at Month 7 | 0.04 (0.07) | 0.06 (0.07)
  Change From Baseline at Month 8: number analyzed (Participants) | 38 | 34
  Change From Baseline at Month 8 | 0.05 (0.08) | 0.07 (0.07)
  Change From Baseline at Month 9: number analyzed (Participants) | 38 | 35
  Change From Baseline at Month 9 | 0.07 (0.11) | 0.09 (0.13)
  Change From Baseline at Month 10: number analyzed (Participants) | 37 | 34
  Change From Baseline at Month 10 | 0.06 (0.07) | 0.06 (0.07)
  Change From Baseline at Month 11: number analyzed (Participants) | 38 | 32
  Change From Baseline at Month 11 | 0.05 (0.07) | 0.08 (0.08)
  Change From Baseline at Month 12: number analyzed (Participants) | 36 | 36
  Change From Baseline at Month 12 | 0.06 (0.12) | 0.07 (0.08)
  Change From Baseline at Month 13: number analyzed (Participants) | 34 | 34
  Change From Baseline at Month 13 | 0.04 (0.08) | 0.08 (0.08)
  Change From Baseline at Month 14: number analyzed (Participants) | 33 | 31
  Change From Baseline at Month 14 | 0.08 (0.07) | 0.08 (0.08)
  Change From Baseline at Month 15: number analyzed (Participants) | 37 | 30
  Change From Baseline at Month 15 | 0.06 (0.07) | 0.06 (0.08)
  Change From Baseline at Month 16: number analyzed (Participants) | 36 | 29
  Change From Baseline at Month 16 | 0.05 (0.08) | 0.08 (0.09)
  Change From Baseline at Month 17: number analyzed (Participants) | 33 | 27
  Change From Baseline at Month 17 | 0.07 (0.08) | 0.08 (0.09)
  Change From Baseline at Month 18: number analyzed (Participants) | 30 | 27
  Change From Baseline at Month 18 | 0.05 (0.09) | 0.09 (0.07)
  Change From Baseline at Month 19: number analyzed (Participants) | 29 | 25
  Change From Baseline at Month 19 | 0.06 (0.10) | 0.09 (0.10)
  Change From Baseline at Month 20: number analyzed (Participants) | 27 | 20
  Change From Baseline at Month 20 | 0.04 (0.08) | 0.11 (0.08)
  Change From Baseline at Month 21: number analyzed (Participants) | 27 | 23
  Change From Baseline at Month 21 | 0.09 (0.12) | 0.09 (0.10)
  Change From Baseline at Month 22: number analyzed (Participants) | 29 | 23
  Change From Baseline at Month 22 | 0.06 (0.08) | 0.09 (0.10)
  Change From Baseline at Month 23: number analyzed (Participants) | 25 | 24
  Change From Baseline at Month 23 | 0.07 (0.06) | 0.12 (0.08)
  Change From Baseline at Month 24: number analyzed (Participants) | 34 | 31
  Change From Baseline at Month 24 | 0.07 (0.08) | 0.12 (0.10)
  Change From Baseline at Follow Up Day 7: number analyzed (Participants) | 2 | 7
  Change From Baseline at Follow Up Day 7 | -0.01 (0.02) | 0.14 (0.08)
  Change From Baseline at End of Treatment: number analyzed (Participants) | 5 | 7
  Change From Baseline at End of Treatment | -0.01 (0.11) | 0.02 (0.08)
  Change From Baseline at Last Visit | 0.05 (0.09) | 0.10 (0.08)

20. Secondary Outcome: Phase A and B: Percentage of Participants With Potentially Clinically Significant Abnormalities in Vital Signs
Description: Vital sign measurements included measurements of respiratory rate, blood pressure, body temperature and pulse. Any value outside the normal range was flagged for the attention of the investigator who assessed whether or not a flagged value is of clinical significance. Only those categories with at least one participant with event are reported. As prespecified in the protocol, data for safety is reported by the treatment group (Phase A: Tolvaptan, Phase A: Placebo, Phase B: Prior Tolvaptan and Phase B: Prior Placebo).
Time Frame: From first dose of study drug up to 14 days post last dose (up to approximately 37 months)
Population: The Phase A Safety Set included all participants who were randomized and received at least 1 dose of IMP in Phase A. The Phase B Safety Set included all participants who were enrolled in Phase B and received at least 1 dose of IMP in Phase B. Number analyzed is the number of participants with at least one post-baseline numeric result for the given vital sign parameter.
Measure: Number; unit: percentage of participants
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 48 | 43 | 42 | 39
percentage of participants
  Pulse Rate (Beats per Minute [BPM]) <=50 and Decrease from Baseline >=15: number analyzed (Participants) | 48 | 43 | 42 | 38
  Pulse Rate (Beats per Minute [BPM]) <=50 and Decrease from Baseline >=15 | 0.0 | 2.3 | 0.0 | 5.3
  Systolic Blood Pressure (millimetre of mercury [mmHg]) >=130 and Increase from Baseline >=20 | 2.1 | 0.0 | 0.0 | 0.0
  Systolic Blood Pressure (mmHg) <=120 and Decrease from Baseline >=20 | 4.2 | 7.0 | 9.5 | 10.3
  Systolic Blood Pressure (mmHg) >=144 and Increase from Baseline >=20 | 2.1 | 2.3 | 0.0 | 2.6
  Diastolic Blood Pressure (mmHg) <=50 and Decrease from Baseline >=15 | 4.2 | 7.0 | 9.5 | 0.0
  Diastolic Blood Pressure (mmHg) >=86 and Increase from Baseline >=15 | 0.0 | 0.0 | 7.1 | 0.0
  Diastolic Blood Pressure (mmHg) <=80 and Decrease from Baseline >=15 | 12.5 | 18.6 | 16.7 | 12.8
  Diastolic Blood Pressure (mmHg) >=92 and Increase from Baseline >=15 | 0.0 | 4.7 | 4.8 | 2.6

21. Secondary Outcome: Phase A and B: Percentage of Participants With Potentially Clinically Significant Abnormalities in Laboratory Test Results Including Liver Function Tests (LFTs)
Description: Laboratory parameters=haematology,chemistry,urinalysis,& LFTs.Criteria for laboratory abnormalities along with their test result grade=Increased creatinine level: Baseline(BSL):Grade 0,>BSL-1.5xBSL:1,>1.5-3xBSL:2,>3-6xBSL:3,>6xBSL:4.Decreased glucose level: <30:-4,30-<40:-3, 40-<55:-2, 55-<65:-1,>=65:0; Increased:<=115:0,>115-160:1,>160-250:2,>250-500:3,>500:4.Decreased potassium level: <2.5:-4,2.5-<3:-3,3-<lower limit of normal(LLN):-1,LLN:0; Increased:upper limit of normal(ULN):0,>ULN-5.5:1,>5.5-6:2,>6-7:3,>7:4.Decreased sodium level: <120:-4,120-124:-3,125-129:-2,130-135:-1,>=136:0; Increased:<=145:0,146-150:1,151-155:2,156-160:3,>160:4. Increased triglyceride level:ULN:0,>ULN-2.5xULN:1,>2.5-5xULN:2,>5-6xULN:3,>6xULN:4. Decreased Neutrophils:<0.5:-4,0.5-<1:-3,1-<1.5:-2,1.5-<LLN:-1,LLN:0. Potentially clinically significant increase or decrease was defined as Baseline grade 0,1,-1 and post-baseline grade >1, <-1 or Baseline grade >1,<-1 and post-baseline grade >or<Baseline grade.
Time Frame: From first dose of study drug up to 14 days post last dose (up to approximately 37 months)
Population: The Phase A Safety Set included all participants who were randomized and received at least 1 dose of IMP in Phase A. The Phase B Safety Set included all participants who were enrolled in Phase B and received at least 1 dose of IMP in Phase B. Number analyzed is the number of participants with at least one post-baseline numeric result for the given laboratory parameter. Only those categories with at least one participant with event are reported.
Measure: Number; unit: percentage of participants
Groups:
- Phase B: Prior Placebo: Qualified participants (defined as those who were willing to continue in the trial and who did not have any AEs that would require IMP discontinuation) who received matching-placebo and completed Phase A, were enrolled in Phase B and received tolvaptan tablets, orally as a split dose (with the first dose taken upon awakening and the second dose taken approximately 8 hours later), based on their current body weight as per following specifications: ≥20 to <45 kg: 15/7.5 mg; ≥45 to ≤75 kg: 30/15 mg; >75 kg: 45/15 mg, for 1 week. The starting dose was up-titrated (≥20 to <45 kg: 30/15 mg; ≥45 to ≤75 kg: 45/15 mg; >75 kg: 60/30 mg) after 1 week based upon tolerability and thereafter participants continued the same dose for 24 months. Doses may be titrated down dependent upon participant tolerability.
  Period Title: Phase A: Double-blind Period (12 Months)
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 48 | 43 | 42 | 39
percentage of participants
  Increase in Creatinine Level (mg/dL) | 8.3 | 0.0 | 7.1 | 7.7
  Decrease in Glucose Level (mg/dL): number analyzed (Participants) | 36 | 39 | 32 | 34
  Decrease in Glucose Level (mg/dL) | 0.0 | 2.6 | 0.0 | 2.9
  Increase in Potassium Level (milliequivalents per deciliter [mEq/dL]): number analyzed (Participants) | 47 | 43 | 40 | 38
  Increase in Potassium Level (milliequivalents per deciliter [mEq/dL]) | 2.1 | 0.0 | 0.0 | 2.6
  Increase in Sodium Level (mEq/dL) | 0.0 | 0.0 | 0.0 | 2.6
  Increase in Triglyceride Level (mg/dL): number analyzed (Participants) | 36 | 39 | 32 | 34
  Increase in Triglyceride Level (mg/dL) | 0.0 | 0.0 | 3.1 | 0.0
  Decrease in Neutrophils (10^9/L): number analyzed (Participants) | 46 | 41 | 40 | 38
  Decrease in Neutrophils (10^9/L) | 0.0 | 4.9 | 5.0 | 2.6

22. Secondary Outcome: Phase A and B: Percentage of Participants With Aquaretic Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. Aquaretic AEs included Medical Dictionary for Regulatory Activities [MedDRA] preferred terms of thirst, polyuria (production of large volumes of dilute urine), nocturia (need to wake up to urinate at night), pollakiuria (abnormally frequent urination), and polydipsia (excessive thirst). As prespecified in the protocol, data for safety is reported by the treatment group (Phase A: Tolvaptan, Phase A: Placebo, Phase B: Prior Tolvaptan and Phase B: Prior Placebo).
Time Frame: From first dose of study drug up to 14 days post last dose (up to approximately 37 months)
Population: The Phase A Safety Set included all participants who were randomized and received at least 1 dose of IMP in Phase A. The Phase B Safety Set included all participants who were enrolled in Phase B and received at least 1 dose of IMP in Phase B.
Measure: Number; unit: percentage of participants
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
Number analyzed (Participants) | 48 | 43 | 42 | 39
percentage of participants | 64.6 | 16.3 | 14.3 | 48.7

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 14 days post last dose (up to approximately 37 months)
Description: The Phase A Safety Set included all participants who were randomized and received at least 1 dose of IMP in Phase A. The Phase B Safety Set included all participants who were enrolled in Phase B and received at least 1 dose of IMP in Phase B. As prespecified in the protocol, data for safety is reported by the treatment group (Phase A: Tolvaptan, Phase A: Placebo, Phase B: Prior Tolvaptan and Phase B: Prior Placebo).
Arm/Group | Phase A: Tolvaptan | Phase A: Placebo | Phase B: Prior Tolvaptan | Phase B: Prior Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/43 | 0/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/48 | 6/43 | 7/42 | 8/39
Other Adverse Events (participants affected / at risk) | 45/48 | 42/43 | 38/42 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A: Tolvaptan (N=48) | Phase A: Placebo (N=43) | Phase B: Prior Tolvaptan (N=42) | Phase B: Prior Placebo (N=39)
Viral pericarditis (Infections and infestations) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Petit mal epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal pain (Renal and urinary disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 2 | 0
Expired product administered (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2
Heart rate increased (Investigations) | 0 | 0 | 0 | 1
SARS-COV-2 test positive (Investigations) | 0 | 0 | 1 | 1
Eating disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase A: Tolvaptan (N=48) | Phase A: Placebo (N=43) | Phase B: Prior Tolvaptan (N=42) | Phase B: Prior Placebo (N=39)
Ear pain (Ear and labyrinth disorders) | 3 | 2 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 3 | 4 | 12
Abdominal pain upper (Gastrointestinal disorders) | 5 | 4 | 5 | 4
Constipation (Gastrointestinal disorders) | 5 | 1 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 3 | 5
Nausea (Gastrointestinal disorders) | 3 | 7 | 7 | 5
Vomiting (Gastrointestinal disorders) | 7 | 10 | 5 | 7
Asthenia (General disorders) | 0 | 3 | 3 | 2
Fatigue (General disorders) | 4 | 3 | 3 | 3
Pyrexia (General disorders) | 4 | 3 | 8 | 7
Thirst (General disorders) | 7 | 2 | 1 | 3
Seasonal allergy (Immune system disorders) | 4 | 1 | 0 | 3
Bronchitis (Infections and infestations) | 3 | 1 | 2 | 2
Ear infection (Infections and infestations) | 1 | 4 | 3 | 2
Nasopharyngitis (Infections and infestations) | 10 | 14 | 11 | 13
Pharyngitis (Infections and infestations) | 4 | 0 | 3 | 2
Rhinitis (Infections and infestations) | 3 | 3 | 11 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 2 | 2 | 5
Viral infection (Infections and infestations) | 3 | 1 | 5 | 3
Blood creatinine increased (Investigations) | 9 | 2 | 7 | 5
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1 | 5
Polydipsia (Metabolism and nutrition disorders) | 5 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 6 | 1 | 3
Dizziness (Nervous system disorders) | 3 | 5 | 4 | 4
Headache (Nervous system disorders) | 16 | 21 | 15 | 17
Migraine (Nervous system disorders) | 2 | 3 | 1 | 2
Nocturia (Renal and urinary disorders) | 7 | 3 | 1 | 6
Pollakiuria (Renal and urinary disorders) | 9 | 0 | 1 | 2
Polyuria (Renal and urinary disorders) | 13 | 2 | 2 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 7 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 9 | 7
Hypertension (Vascular disorders) | 4 | 1 | 4 | 2
Orthostatic hypotension (Vascular disorders) | 5 | 0 | 3 | 3
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 3 | 0
Cystitis (Infections and infestations) | 0 | 0 | 3 | 0
Gastoenteritis (Infections and infestations) | 0 | 0 | 3 | 5
Sinusitis (Infections and infestations) | 0 | 0 | 3 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 4 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Viral upper respiratory tractinfection (Infections and infestations) | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 3
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2
Liver function test increased (Investigations) | 0 | 0 | 0 | 2
Vitamin D decreased (Investigations) | 0 | 0 | 4 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Enuresis (Psychiatric disorders) | 0 | 0 | 2 | 2
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 3
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 3
Renal pain (Renal and urinary disorders) | 0 | 0 | 4 | 3
Hypotension (Vascular disorders) | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT02964273/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT02964273/SAP_001.pdf